CLINICAL TRIAL: NCT06772285
Title: Single Arm Feasibility Study of a Digital Health App to Support Adults With Managing a PEG Feeding Tube After Insertion
Brief Title: Albert Health App PEG Study
Acronym: Albert
Status: Not yet recruiting | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024GAS132
Record Dates: First submitted 2025-01-02; First posted 2025-01-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Feeding Tube Complication
Keywords: Digital health app; Management; PEG; Feeding tube; Insertion; Albert Health; PEG insertion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PEG tube electively inserted: Adults ≥18 years and/or the carer of a person ≥18 having a PEG tube electively inserted
  Interventions: Other: Albert Health app

INTERVENTIONS:
Other: Albert Health app — Test an existing digital health app, called Albert Health, designed to support patients with a newly inserted feeding tube to use and manage their tube care, in a feasibility study.

SUMMARY:
Test an existing digital health app, called Albert Health, designed to support patients with a newly inserted feeding tube to use and manage their tube care, in a feasibility study. The feasibility study will evaluate the acceptability, usability and accessibility of the app in preparation for a randomised controlled trial.

DETAILED DESCRIPTION:
Seven thousand people have a feeding tube inserted directly into the stomach or bowel in the UK each year for the purposes of giving fluid, food or medication via the tube instead of orally. Over one third will experience a complication in the first 12 months after insertion, half of whom will experience it in the first 30 days. For the majority of people pain, infection and leaking are the commonest early complications; for most, these complications are minor and do not require intervention. But they also mimic the symptoms of more serious complications, making it an anxious time for patients and carers and hard for them to discern if and what level of help they need. Six percent of all people with a PEG will have to spend time in hospital having the problem investigated or managed and 5% will die in the first 30 days after a tube insertion, predominantly from procedure related complications.

Currently the insertion of a feeding tube is an invasive process, undertaken on both inpatients and outpatients for a variety of medical reasons including the need for cancer treatment and for medium- or long-term neurological conditions and/or severe learning disabilities (LD) affecting swallowing, often with multiple comorbidities. All these populations have a higher mortality, and in this situation are often further disadvantaged by their illness affecting their ability to communicate. The LD population in particular suffer from inequities of healthcare outcomes and are underrepresented in the physical health research arena.

After the procedure and discharge people/carers are supported by a multidisciplinary team, including a community nurse, to help them use their tube and the associated equipment and information to troubleshoot tube problems in accordance with NICE guidance. This includes use of a pharma-owned digital app for simple device guidance around the electronic equipment. Some areas in the UK have nutrition nurse specialist teams that can be contacted during weekdays for support.

Should a significant complication occur out of normal working hours, people with feeding tubes often end up attending the emergency department as they do not have access to support or advice. This is common as people tend to use their tubes in the evening.

Patients and family in the investigators Patient Advisory Group (PAG) reported it was an 'overwhelming' and 'frightening' experience living with a PEG tube in the first few weeks. The group reported it was hard to access support as an outpatient and slow response to support requests led to unnecessary admissions or prolonged hospital stays. There was a perception of a lack of transition of care between the hospital and community setting and better or repeated information earlier in the process could reduce the learning curve of how to manage their feeding tubes. The group described that, currently provided, written information in the form of leaflets was perceived as "very daunting" and a "bit scary at first". The group suggested the investigators focus on improving the support around implementing the training they received in hospital and access to early advice. All patients reported they used the pharma company apps and would be willing to use an app to support them or ease the transition phase from secondary to community care.

In the event people with feeding tubes attend the emergency department, there is often not a need for admission, and they can be managed with simple advice or measures, and these are preventable attendances. Where rapid care is required to prevent admission, delays to care can result in avoidable admissions and our PPI group expressed frustration that this was occurring when it could be prevented with better access to advice or support.

Albert Health is a digital app used in Turkey, where it is nationally commissioned to support >6000 professional carers with enteral feeding tubes to manage simple problems for themselves and know when to access help. In the UK over half of our patients manage their feeding tubes themselves or within their nuclear families.

Therefore, the investigators have an underserved population identifying a specific need for support, who suffer healthcare inequalities and have healthcare accessibility challenges, but who the investigators know will, and do, use app technology for tube management. The investigators propose to employ a successful and internationally utilised app, with content co-designed and created with PPI to offer that additional support and advice to improve the health and wellbeing of our people with newly inserted feeding tubes. A secondary effect will be reducing the burden on the healthcare system and tackling healthcare inequalities in a multi-morbid population.

The investigators have created English language versions of the content that adheres to UK guidance, that is accessible by voice access and by typing and touch screen. The content and 'nudges' have been co-created with patients and carers to be suitable for patients themselves and their familial carers and both content and nudges are tube-type specific to offer them a personalised experience. The app uses nudge technology to highlight key dates after tube insertion for specific care and support and answers commonly asked questions, with supportive subtitled video content on using the tube, looking after the tube and dealing with simple problems. The app also allows users to set reminders to help maintain good care of the tube over the longer term, which will help prevent longer-term serious complications.

This feasibility study would test the app in the UK and understand if the adapted version works as intended as an intervention, if it is acceptable to patients, if it is useable and accessible, and if this population would be readily recruited to a larger research study. Answering these questions would determine if the app would be suitable to be tested in a randomised controlled trial against standard care and collate data to define the parameters of that future study. This clinical population are often disabled, and this will allow us to focus on if the accessibility adaptations are suitable and if it is usable in the intended population and if recruitment amongst this population to support a larger study is feasible.

Percutaneous endoscopic gastrostomy (PEG), a technique first described in 1980 provides long-term enteral nutrition access in patients with a functional gastrointestinal tract and impaired swallowing. PEGs are better tolerated and associated with better nutritional outcomes and fewer complications than nasogastric tubes and therefore guidelines recommend PEG for prolonged enteral supplementation.

PEG insertion is invasive; complications can include bowel perforation, bleeding, infection and tube displacement. The 2004 National Confidential Enquiry into Patient Outcome and Death report reviewed all UK deaths associated with PEG procedure between April 2002 and March 2003. The report found that 20% of PEGs were futile or not indicated, 40% had concurrent chest infection and 43% of deaths occurred within 7 days of the procedures. A follow up population-based study in the UK has demonstrated improved patient outcomes at a national level with a reduction in all-cause 30 day mortality of 60% following PEG insertion between 2007 and 2019.

A recent UK national report highlighted substantial variation in 30-day mortality rates following PEG insertion. One possible reason suggested was variation in nutrition support team provision across the UK, 16.7% of providers have no nutrition support and 25% no dedicated nutrition nurse specialist.

Experiencing complications is common. In a single-centre UK study between 2016-2018, 80% of PEG recipients were cared for in their own home and 16.7% experienced a complication in the first 30 days, with over 35% having a complication within 12 months. The most common complication was pain, for which home-cared patients were more likely to seek medical attention than patients from nursing homes. In a study by Barret et al 2021 identified that an Emergency Department attendance for a PEG tube problem cost an average of $1061 per person manifested in days in hospital and procedural costs, as well as patient morbidity with over half of the ED attendances resolved at the bedside.

Qualitative studies on patients experience with a PEG tube identified challenges adapting both physically and psychosocially. Discomfort was commonly described, and much effort and time was spent managing tube problems, often without support from knowledgeable healthcare professionals. Additionally, people with enteral tubes needed considerable support from knowledgeable, responsive healthcare professionals during the weeks following initial placement of the enteral tube, leading them to recommend 24-hour services designed in partnership with patients to support, reduce burden, negative experience, waste and hospital admissions.

Therefore, the investigators have a predominantly home-based population with enteral tubes, likely to experience pain and challenges, especially shortly after PEG insertion, that would prompt them to seek medical reassurance and support without requiring an inpatient admission. This occurs in a country with a geographically variable hospital-based nutrition support service and in a disease-specific population familiar with app-based technology as part of the standard care in the UK.

The Albert Health app aims to meet that need using an advanced digital healthcare app that is already successful for this purpose, utilised and nationally commissioned in an EU country. It has been redesigned in partnership with UK patients, public and healthcare staff to offer practical support, reassurance, signposting, education and behavioural modification to reduce negative experience and burden on patients at home with an enteral tube and ultimately reduce attendances at hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Person ≥18 and/or the carer of a person ≥18 having a PEG tube electively inserted; the participant or their supporting carer must be literate in English.
2. Written informed consent for study participation obtained from the patient or personal consultee (friend/family), with assent as appropriate by the patient, depending on the level of understanding.

   a. Where a personal consultee is the primary participant (ie user of the app) it must be understood that data will be required and collected on the person they are supporting with the app and PEG tube.
3. Willingness to comply with all study requirements.
4. The participant or carer must have access to a smart phone or mobile device (such as a pad).

Exclusion Criteria:

1. Person being discharged to a nursing home
2. Both participant and carer are visually impaired.
3. Patient's whose PEG care will be solely provided by district nurses or professional health care workers
4. Patient has major surgery scheduled within 7 days of the PEG insertion date

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients (adults) seen at New Cross Hospital or City Sandwell Hospital undergoing an elective percutaneous endoscopic gastrostomy will be approached. Participants may be recruited in the following partnerships:
  i) Primary app user is patient, who will be self-caring, willing to take part and able to consent ii) Co-primary app - patient and carer, both willing to take part and sharing the tube care and able to consent iii) Primary app user is carer providing most or all tube care, willing to take part, carer consent
  1. Patient willing to consent - patient consent
  2. Patient unable to consent- consultee consent
  There is no upper age limit for participation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the acceptability of the app intervention to users | Day 14 and 28
  Evaluate the acceptability of the app intervention to users ; interviews, MARS day 14 and 28
Evaluate the useability and interaction with the app by users | 18 months
  Evaluate the useability and interaction with the app by users ; interviews, internal app measures
Evaluate the accessibility of the app to users | 18 months
  Evaluate the accessibility of the app to users ; interviews
Evaluate the accessibility of the app to users | 18 months
  Evaluate the accessibility of the app to users ; satisfaction scores (SUS subcale)
Evaluate the accessibility of the app to users | 18 months
  Evaluate the accessibility of the app to users ; MAUQ-E subscales
Evaluate the useability and interaction with the app by users | Day 21
  Evaluate the useability and interaction with the app by users ; System Usability Scale SUS
Evaluate the useability and interaction with the app by users | Day 21
  Evaluate the useability and interaction with the app by users ; MAUQ-E
Evaluate ability to recruit this specific patient and carer population into a research trial | 18 months
  Evaluate ability to recruit this specific patient and carer population into a research trial ; recruitment rate
Evaluate ability to recruit this specific patient and carer population into a research trial | 18 months
  Evaluate ability to recruit this specific patient and carer population into a research trial ; numbers approached versus numbers recruited
Evaluate ability to recruit this specific patient and carer population into a research trial | 18 months
  Evaluate ability to recruit this specific patient and carer population into a research trial ; percentage who complete the study period
Evaluate ability to recruit this specific patient and carer population into a research trial | 18 months
  Evaluate ability to recruit this specific patient and carer population into a research trial ; questionnaire completion rates

CONTACTS AND LOCATIONS:
Overall Officials: Helen Steed, Principal Investigator — Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom